CLINICAL TRIAL: NCT00058968
Title: Duloxetine Versus Placebo in the Treatment of Patients With Painful Diabetic Neuropathy
Brief Title: A Study for the Treatment of Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4097; F1J-MC-HMAV
Record Dates: First submitted 2003-04-15; First posted 2003-04-16 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Diabetic Neuropathy, Painful
Keywords: neuropathy; pain; diabetes; chronic pain; persistent pain; leg pain; peripheral neuropathy; foot pain; painful neuropathy; diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Diabetes Mellitus; Chronic Pain; Peripheral Nervous System Diseases; Neuropathy, Painful | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine hydrochloride
Drug: placebo

SUMMARY:
The purpose of the study is to determine if duloxetine can help patients with painful diabetic neuropathy.

DETAILED DESCRIPTION:
The protocol will assess the efficacy and safety of duloxetine. It will also look at how duloxetine affects quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age.
* Patients with pain due to diabetic neuropathy in both legs.
* Females must not be pregnant or plan to become pregnant during the study.
* Stable Glycemic control.
* Average mean pain severity score of at least 4.0 as assessed by completion of a daily diary.

Exclusion Criteria:

* You are related to or work for the physician conducting the study or are employed by Eli Lilly and Company.
* You have a severe or serious medical condition that causes you to be hospitalized often; or you have had a kidney transplant or are on current dialysis.
* You have participated in a study for an investigational drug within the last 30 days.
* You have a history of major depressive disorder, generalized anxiety disorder, or alcohol or eating disorders.
* You have a past medical history or diagnosis of mania, bipolar disorder, or psychosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660
Dates: Start 2002-10; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Reduction in average pain severity as measured by an 11-point Likert scale.

SECONDARY OUTCOMES:
Pain severity for worst pain and night pain as measured by an 11-point Likert scale.
Clinical Global Impression of Severity scale to measure severity of illness at the time of assessment.
Patient Global Impression of Improvement scale to measure the degree of improvement at the time of assessment.
Brief Pain Inventory to measure the severity of pain.
Sensory Portion of the Short Form McGill pain questionnaire measures severity of 11 pain descriptors.
Hamilton Depression Rating Scale (17 item) used to assess severity of depression symptoms during the course of therapy.
Dynamic Allodynia measure to elicit the pain severity to a normally non-painful stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLilly (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida, United States

REFERENCES:
- [Derived] Ziegler D, Pritchett YL, Wang F, Desaiah D, Robinson MJ, Hall JA, Chappell AS. Impact of disease characteristics on the efficacy of duloxetine in diabetic peripheral neuropathic pain. Diabetes Care. 2007 Mar;30(3):664-9. doi: 10.2337/dc06-2009. PMID 17327338
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com